CLINICAL TRIAL: NCT02360345
Title: A Phase I Trial of ONX-0801 (a Novel α-folate Receptor-mediated Thymidylate Synthase Inhibitor) Exploring Once Weekly and Alternate Week Dosing Regimens in Patients With Solid Tumours
Brief Title: Phase I Trial of ONX-0801 Once Weekly or Alternate Weekly
Acronym: ONX-0801
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR3941; 2013-000569-34 (EudraCT Number)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumours
MeSH Terms: interventions — BGC945

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- q1week schedule (Experimental): ONX-0801 will be administered over a 1-hour IV infusion on Days 1, 8, 15 and 22 of repeated 28-day treatment cycles.
  Interventions: Drug: ONX-0801
- q2week schedule (Experimental): ONX-0801 will be administered over a 1-hour IV infusion on Days 1 and 15 of repeated 28-day treatment cycles.
  Interventions: Drug: ONX-0801

INTERVENTIONS:
Drug: ONX-0801

SUMMARY:
This is an open label, single-centre dose escalation phase 1 clinical trial of ONX-0801.

The study will evaluate two schedules of ONX-0801 concurrently: once weekly and alternate week dosing, of repeated 28-day treatment cycles.

The study will consist of two stages: the dose escalation phase, in which the recommended phase II dose will be determined; and the expansion phase, in which up to 30 patients will be treated at the recommended phase II dose and schedule to further support the design of subsequent trials of ONX-0801.

DETAILED DESCRIPTION:
During the dose escalation phase, patients will be enrolled alternately to either:

* a q1wk schedule in which ONX-0801 will be administered over a 1-hour IV infusion on Days 1, 8, 15 and 22 of repeated 28-day treatment cycles; the starting dose will be 1 mg/m2 for the first cohort; OR
* a q2wk schedule in which ONX-0801 will be administered over a 1-hour IV infusion on Days 1 and 15 of repeated 28-day treatment cycles; the starting dose will be 2 mg/m2 for the first cohort;

Cohorts of 3 patients will receive ONX-0801 at escalating doses on each schedule until a Dose Limiting Toxicities (DLTs) occur and an Maximum Tolerated Dose (MTD) is determined for each schedule.

Once the recommended Phase II dose (RP2D) and schedule has been established, additional patients may be recruited in a dose expansion phase to a maximum total of 30 patients to further characterize safety, tolerability and pharmacodynamics. This subgroup of patients will be limited to those expected to have high rates of over expression of α-FR, such as patients with ovarian or endometrial, cancer.

Approximately 66 patients with solid tumours will be entered into this study.

Dose escalation: Approximately 18 patients in each schedule in the dose escalation phase. The final number for the dose escalation phase will depend on the number of dose escalations required to reach DLT.

Dose expansion: Up to 30 patients will be enrolled in the dose expansion phase, and this cohort will be enriched with patients with tumour types expected to have high rates of over expression of α-folate receptor, including ovarian and endometrial cancer. A minimum of 20 patients with platinum resistant/refractory ovarian cancer will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven solid tumours (to include Non-Hodgkin's and Hodgkin's lymphoma). Patients must have disease which has failed standard therapy or for whom no standard curative therapy exists. At the dose expansion phase, entry will be limited to patients with ovarian and endometrial cancers with availability of archival paraffin embedded tissue
* Measurable (as defined by RECIST version 1.1) or evaluable (based on tumour markers) disease
* Life expectancy of at least 12 weeks
* World Health Organisation (WHO) performance status of 0-1 (Appendix 1)
* Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.

Laboratory Test Value required Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible Serum creatinine ≤ 1.5 x ULN PT and APTT ≤ 1.25x ULN

* Normal (no clinically significant abnormalities) 12-lead ECG, QTc interval <470 ms
* Pulmonary function test FVC of >70%, DLCOc (DLCO corrected for Hb) of >60%
* 18 years or over
* Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

Exclusion Criteria:

* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and 4 weeks for investigational medicinal products) before treatment.
* Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDU should not exclude the patient
* Patients with new brain metastases. Patients with treated (surgically excised or irradiated) and stable brain metastases are eligible as long as the treatment was at least 4 weeks prior to initiation of study drug and brain MRI within 2 weeks of initiation of study drug is negative for new metastases.
* Patients with pulmonary metastases
* History of thoracic radiation or other history likely to create pre-existing lung disease
* Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have a intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible..
* Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
* Major thoracic or abdominal surgery from which the patient has not yet recovered.
* Patients with sub-acute bowel obstruction
* Patients using heparin, or warfarin/coumadin type anticoagulants, however, low-dose (<2mg) coumadin for portacath patency is allowed;
* Organ transplant recipients
* Patients with known systemic disease with pulmonary involvement, including active uncontrolled infection.
* Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Patients with history of QT prolongation, clinically significant VT, VF, heart block, MI within 1 year, CHF NYHA Class III or IV, unstable angina, angina within 6 months, or other evidence of clinically significant coronary artery disease
* Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of ONX-0801. Participation in an observational trial would be acceptable.
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 cycles (56 days)
  Establish the maximum tolerated dose of ONX-0801 when given on a weekly or alternate weekly schedule.
Safety and Toxicity Profile 9adverse event to ONX-0801 and grading severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0) | 2 cycles (56 days)
  Assign causality of each adverse event to ONX-0801 and grading severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

SECONDARY OUTCOMES:
Pharmacokinetic profile of ONX-0801 (Cmax, AUC and volume of distribution) | 36 months
  Document Cmax, AUC and volume of distribution of ONX-0801 and determine if it is possible to achieve a plasma concentration of ≥ 0.05μM at the maximally tolerated dose in each schedule.

OTHER OUTCOMES:
Anti-tumour activity (disease response by RECIST criteria version 1.1) | 36 months
  Determine disease response by RECIST criteria version 1.1, GCIC CA125 criteria and change in tumour size.
Predictive Biomarkers (Analyse archival tumour tissue for α-FR) | 36 months
  Analyse archival tumour tissue for α-FR as a predictive biomarker of disease response to ONX-0801. Correlate anti-tumour activity with the expression of α-FR
Pharmacodynamic behaviour of ONX-0801 (levels of apoptosis markers (m30 and m65) in surrogate tissue) | 36 months
  To determine the levels of apoptosis markers (m30 and m65) in surrogate tissue

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, MBBS, PhD, Principal Investigator — The Institute of Cancer Research, The Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Result] Banerjee S, Michalarea V, Ang JE, Ingles Garces A, Biondo A, Funingana IG, Little M, Ruddle R, Raynaud F, Riisnaes R, Gurel B, Chua S, Tunariu N, Porter JC, Prout T, Parmar M, Zachariou A, Turner A, Jenkins B, McIntosh S, Ainscow E, Minchom A, Lopez J, de Bono J, Jones R, Hall E, Cook N, Basu B, Banerji U. A Phase I Trial of CT900, a Novel alpha-Folate Receptor-Mediated Thymidylate Synthase Inhibitor, in Patients with Solid Tumors with Expansion Cohorts in Patients with High-Grade Serous Ovarian Cancer. Clin Cancer Res. 2022 Nov 1;28(21):4634-4641. doi: 10.1158/1078-0432.CCR-22-1268. PMID 35984704